CLINICAL TRIAL: NCT01586117
Title: A Phase II Study of Amifostine for the Prevention of Acute Radiation-Induced Rectal Toxicity
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Jin, M.D., M.D. Cancer Hospital, CAMS, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CH-GI-022
Record Dates: First submitted 2012-04-22; First posted 2012-04-26 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; amifostine; pre-operative chemo-radiation
MeSH Terms: conditions — Rectal Neoplasms | interventions — Amifostine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Amifostine (Experimental): intrarectal Amifostine assign to the Amifostine arm
  Interventions: Drug: Amifostine

INTERVENTIONS:
Drug: Amifostine — intrarectal Amifostine administration 1500mg QD x 5 weeks

SUMMARY:
The purpose of this study is to evaluate the effect of intrarectal Amifostine administration on acute radiation-induced rectal toxicity in pre-operative chemo-radiotherapy.

DETAILED DESCRIPTION:
To evaluate the different use way of intrarectal Amifostine administration on acute radiation-induced rectal toxicity in pre-operative chemo-radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed rectal cancer, preoperative stage II / III (T3-4N0 or T1-4N + M0).
* tumor distance from anus less than 12 cm.
* KPS score not less than 70
* can be tolerated chemotherapy and radiotherapy.
* pelvic who had no history of radiation therapy.
* Non-allergic history of fluorouracil or platinum-based chemotherapy drugs.
* blood pressure can be controlled by drugs in the normal range (90 ≤ systolic blood pressure ≤ 140,60 ≤ diastolic blood pressure ≤ 90).
* a full understanding of the study, the ability to complete all of the treatment plan, follow up the conditions and sign the informed consent.

Exclusion Criteria:

* other malignancy (past or at the same time), does not include curable non-melanoma skin cancer and cervical carcinoma in situ; does not include resectable primary colon cancer (synchronous or metachronous).
* pregnant or lactating patients.
* fertility but did not use contraceptive measures.
* existing active infection.
* merge serious complications, can not tolerate the treatment, such as 6 months of myocardial infarction, mental illness, uncontrollable diabetes or uncontrollable hypertension or hypotension.
* concurrent treatment with other anticancer drugs.
* can not complete treatment or follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Acute radiation-induced toxicity: daily diarrhea frequency | about 3 months from chemo-raditherapy to operation

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jin, M.D, Principal Investigator — Chinese Acedemy of Medical Scinences
Locations (1):
- Radiation Oncology Depratment, Cancer Hospital, CAMS, Beijing, Beijing Municipality, China